CLINICAL TRIAL: NCT04055805
Title: Health and Quality of Life in Oncological Patients: Management of Bone Pathology in the Italian Citbl (Cancer Treatment Induced Bone Loss) Population
Brief Title: Health and QoL in Oncological Patients: Management of Bone Pathology in Italian Citbl Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr.ssa Paola Villa, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: VIL-HEQ-17-014
Record Dates: First submitted 2019-03-11; First posted 2019-08-14 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer Female; Osteoporosis
Keywords: Aromatase Inhibitors; Bone pathology; QoL
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Fondazione Policlinico Universitario A. Gemelli, Roma: Polo Scienze della Salute della Donna e del Bambino
  Interventions: Behavioral: Observational Analysis
- Università degli Studi di Pavia
  Interventions: Behavioral: Observational Analysis
- Università di Napoli "Federico II"
  Interventions: Behavioral: Observational Analysis
- Università degli Studi di Siena
  Interventions: Behavioral: Observational Analysis
- Azienda Ospedaliero-Universitaria Careggi Firenze
  Interventions: Behavioral: Observational Analysis
- Fondazione Policlinico Universitario A. Gemelli Roma: U.O.C Chirurgia Senologica
  Interventions: Behavioral: Observational Analysis
- Istituto Nazionale dei Tumori di Napoli Fondazione G.Pascale
  Interventions: Behavioral: Observational Analysis

INTERVENTIONS:
Behavioral: Observational Analysis — Studying the current state of the clinical approaches to bone diseases in breast cancer patients treated with adjuvant and/or hormone therapy

SUMMARY:
Studying the current state of the clinical approaches to bone diseases in breast cancer patients treated with adjuvant and/or hormone therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to provide the Informed consent to participate to the study
* Women aged 18-75 years
* Patients having breast cancer, with no phenotype restrictions
* Patients in natural and stable menopause
* Patients having secondary amenorrhea, that arose after the initiation of oncologic treatment, since at least 12 months or 6 months with FSH> 40 U/I

Exclusion Criteria:

* Patients with advanced cancer and/or bone metastases and/or visceral metastases
* Patients with severe renal insufficiency and/or in dialysis and patients affected by severe endocrine disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: Women affected by breast cancer in menopause or with secondary amenorrhea arising from the initiation of oncologic treatments
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-12-26 (Estimated); Study Completion 2021-10-26 (Estimated)

PRIMARY OUTCOMES:
Results from some questionnaires related to patients QoL, rated from 1 to 10. | 26-32 months
  Description of the current state of the most frequent clinical and therapeutical approaches to bone diseases in 700 breast cancer menopausal patients treated with adjuvant and/or hormonal therapy. These patients are assessed by questionnaires regarding quality of life, menopausal status and current anti resorptive treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Agostino Gemelli, Roma, RM, Italy